CLINICAL TRIAL: NCT04305093
Title: Precision Analytical Retrospective Data Correlation
Brief Title: Data Mining: Precision Analytical Retrospective Data Correlation
Status: Completed | Type: Observational
Sponsor: Precision Analytical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MN11819
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Endocrine; Hormone Disturbance
Keywords: Cortisol; Cortisol metabolites; Obesity; testosterone; estradiol; Hormone therapy; Sleep disturbance; Aging
MeSH Terms: conditions — Obesity; Endocrine System Diseases; Parasomnias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Precision Analytical patients: Individuals who had laboratory work completed at Precision Analytical and completed the associated questionnaire on symptoms and comorbidities.

SUMMARY:
Data from previously analyzed clinical samples tested by Precision Analytical, Inc. will be mined to identify and select samples from patients reporting hormone supplement use. Patient demographics (BMI, for example), different therapies and expected changes in hormone levels will be analyzed and hormone metabolite patterns will be compared. Samples will be deidentified prior to analysis.

DETAILED DESCRIPTION:
The investigators have a list of 10 estrogen metabolites, 8 androgen metabolites, two progesterone metabolites, 4 cortisol metabolites, free cortisol, six organic acids, 8-hydroxy-2'-deoxyguanosine (8-OHdG), and melatonin that are measured on patient urine samples and cortisol and cortisone on patient saliva samples. The investigators would like to both reinforce the validation of the accuracy of these urinary markers and examine how these markers associate with patient demographics, symptoms, hormone therapy doses and routes of administration.

This study will involve analysis of existing data from routine clinical care. All data will be deidentified and each set of results will be given a study ID number. The key will be held by Danielle Martinot and will contain only the original Precision Analytical sample accession number and the new study ID (identification). No identifying PHI (Protected Health Information) will be accessible to the PI.

These data will be used to evaluate the following hypotheses: 1) Urinary hormone measures accurately reflect expected changes in hormones with regard to circadian rhythm, menstrual status, and use of hormonal medications; 2) Urinary metabolites of cortisol will show a stronger association with body mass index and symptoms related to cortisol production as compared to salivary measures; 3) Urine values of reproductive hormones and organic acids will correlate to the dosing of estrogen and androgens more strongly than to progesterone creams; 4) 8-OHdG, a measure of oxidative stress, and melatonin will be correlated with age and BMI; and 5) Urinary hormone measures will capture age-related changes in hormone regulation.

ELIGIBILITY:
Inclusion Criteria:

* Had testing done at Precision Analytical between 2016 and 2019

Exclusion Criteria:

* Varies by data analysis

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 18 and 85 years with data in the Precision Analytical database
Sampling Method: Non-Probability Sample
Enrollment: 144561 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
BMI - weight and height will be combined to report BMI in kg/m2 | 6 months
  Relationship of BMI to cortisol production and clearance
Urinary hormonal profile including concentrations of estrone, estradiol, estriol, alpha-pregnanediol, and beta-pregnanediol | 6 months
  Determination of urine estrogen and progesterone metabolites in postmenopausal women receiving hormonal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Newman, MS, Principal Investigator — Precision Analytical, Inc.
Locations (1):
- Precision Analytical, Inc, McMinnville, Oregon, United States

REFERENCES:
- [Background] Abraham SB, Rubino D, Sinaii N, Ramsey S, Nieman LK. Cortisol, obesity, and the metabolic syndrome: a cross-sectional study of obese subjects and review of the literature. Obesity (Silver Spring). 2013 Jan;21(1):E105-17. doi: 10.1002/oby.20083. PMID 23505190
- [Background] DUNKELMAN SS, FAIRHURST B, PLAGER J, WATERHOUSE C. CORTISOL METABOLISM IN OBESITY. J Clin Endocrinol Metab. 1964 Sep;24:832-41. doi: 10.1210/jcem-24-9-832. No abstract available. PMID 14216471
- [Background] Newman M, Pratt SM, Curran DA, Stanczyk FZ. Evaluating urinary estrogen and progesterone metabolites using dried filter paper samples and gas chromatography with tandem mass spectrometry (GC-MS/MS). BMC Chem. 2019 Feb 4;13(1):20. doi: 10.1186/s13065-019-0539-1. eCollection 2019 Dec. PMID 31384769
- [Background] Pasquali R, Cantobelli S, Casimirri F, Capelli M, Bortoluzzi L, Flamia R, Labate AM, Barbara L. The hypothalamic-pituitary-adrenal axis in obese women with different patterns of body fat distribution. J Clin Endocrinol Metab. 1993 Aug;77(2):341-6. doi: 10.1210/jcem.77.2.8393881.
- [Background] Rask E, Olsson T, Soderberg S, Andrew R, Livingstone DE, Johnson O, Walker BR. Tissue-specific dysregulation of cortisol metabolism in human obesity. J Clin Endocrinol Metab. 2001 Mar;86(3):1418-21. doi: 10.1210/jcem.86.3.7453. PMID 11238541
- [Background] Stimson RH, Andersson J, Andrew R, Redhead DN, Karpe F, Hayes PC, Olsson T, Walker BR. Cortisol release from adipose tissue by 11beta-hydroxysteroid dehydrogenase type 1 in humans. Diabetes. 2009 Jan;58(1):46-53. doi: 10.2337/db08-0969. Epub 2008 Oct 13. PMID 18852329
- [Background] SZENAS P, PATTEE CJ. Studies on adrenocortical function in obesity. J Clin Endocrinol Metab. 1959 Mar;19(3):344-50. doi: 10.1210/jcem-19-3-344. No abstract available. PMID 13631051
- [Background] Tomlinson JW, Finney J, Hughes BA, Hughes SV, Stewart PM. Reduced glucocorticoid production rate, decreased 5alpha-reductase activity, and adipose tissue insulin sensitization after weight loss. Diabetes. 2008 Jun;57(6):1536-43. doi: 10.2337/db08-0094. Epub 2008 Mar 13. PMID 18340018